CLINICAL TRIAL: NCT07108946
Title: Influence of Skin Tone and Background Color on the Accuracy of Auricular Scanning: A Clinical Trial
Brief Title: the Effect of Different Background Color and Skin Tone on the Accuracy of Auricular Scanning
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: yasmine Elsherbeeny (Other)
Responsible Party: Sponsor-Investigator, yasmine Elsherbeeny, lecturer of prosthodontics, faculty of dentistry, ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FDASU-Rec IR032512
Record Dates: First submitted 2025-07-29; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Auricular scan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Type I Fitzpatrick Scale skin tone participant (Experimental): participants of this skin tone will have their ears scanned across three different backgrounds.
  Interventions: Other: Black background; Other: White background; Other: Participant own skin as a background
- Type III Fitzpatrick Scale skin tone participant (Experimental): participants of this skin tone will have their ears scanned across three different backgrounds.
  Interventions: Other: Black background; Other: White background; Other: Participant own skin as a background
- Type IV Fitzpatrick Scale skin tone participant (Experimental): participants of this skin tone will have their ears scanned across three different backgrounds.
  Interventions: Other: Black background; Other: White background; Other: Participant own skin as a background

INTERVENTIONS:
Other: Black background — Changing the background color during scanning to evaluate its effect on scan quality .
Other: White background — Changing the background color during scanning to evaluate its effect on scan quality .
Other: Participant own skin as a background — Changing the background color during scanning to evaluate its effect on scan quality .

SUMMARY:
The goal of this study is to find the best miss and match background color around an ear when taking scans for it , the investigators will recruit participants of three different skin tone and will scan their ear three times; one scan without any background, second scan with black one and the third scan with white background, then the investigators will take an actual physical impression of the participants ear and the investigators will obtain a cast which will be scanned also and its scan will be compared to the three scans taken with different backgrounds to find the best combination.

DETAILED DESCRIPTION:
Manufacturing the Extraoral prosthesis is troublesome for the patient, the dental practitioner and the dental technician. When a person misses his ear congenitally or due to trauma, he wishes to have an accurate replacement for his ear with minimum steps and effort. Digital technology has been providing the dental field with the most helpful equipment in such cases. Owing to the innovation of intraoral scanners with its continuous refinement, this patient now can rest assured that he will have his auricular prosthesis with less number of visits and less effort. There are different environmental factors that can affect scanning accuracy such as patients skin tone and scanning background.This study aims to evaluate the different backgrounds and skin tones effect on the trueness of auricular scanning. Participants with different skin tones (black, white and intermediate) will be selected with intact ears, then conventional impression will be taken and stone cast will be obtained and scanned via an extraoral scanner, then intraoral scanner will be used to scan the auricle three times, first with a black background, second with white background, third without background. Trueness of the scans will be evaluated by metrological software. Data will be collected, tabulated, and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Three types of skin tones will be selected; type I, type III and type VI according to The Fitzpatrick Scale.
2. Participants with intact ears.
3. Participants not exposed to sun burns or tans.

Exclusion Criteria:

* 1- Uncooperative participants.

  * 2-Participants without intact ears.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-07-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of different backgrounds and skin tones on trueness of auricular scans via intraoral scanner. | The study is expected to take place over a 6-week period. Each participant will be scheduled for one session lasting approximately one hour.
  The resultant standard tessellation files (STL) of every scan done via the intraoral scanner will be compared to the STL of the scan done via the extraoral scanner of the same participant by a metrological software to evaluate trueness.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT07108946/Prot_SAP_000.pdf